CLINICAL TRIAL: NCT00369018
Title: Methyl Aminolevulinate (MAL) and Hexaminolevulinate (HAL) Photodynamic Therapy (PDT)of Cervical Intraepithelial Lesions (SIL) - a Double-blind Dose-finding Study
Brief Title: A Dose-finding Study of MAL and HAL Photodynamic Therapy of Cervical Premalignant Lesions.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Photocure (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PC CE101/06
Record Dates: First submitted 2006-08-28; First posted 2006-08-29 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-11

CONDITIONS: Cervical Dysplasia
Keywords: photodynamic therapy; methyl aminolevulinate; hexaminolevulinate; dose-finding; cervical dysplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — methyl 5-aminolevulinate; 5-aminolevulinic acid hexyl ester

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- MAL 3 (Active Comparator)
  Interventions: Drug: methyl aminolevulinate (MAL) and hexaminolevulinate (HAL)
- MAL 12 (Active Comparator)
  Interventions: Drug: methyl aminolevulinate (MAL) and hexaminolevulinate (HAL)
- HAL 10, 3 (Active Comparator)
  Interventions: Drug: methyl aminolevulinate (MAL) and hexaminolevulinate (HAL)
- HAL 10, 12 (Active Comparator)
  Interventions: Drug: methyl aminolevulinate (MAL) and hexaminolevulinate (HAL)
- HAL 40, 3 (Active Comparator)
  Interventions: Drug: methyl aminolevulinate (MAL) and hexaminolevulinate (HAL)
- HAL 40, 12 (Active Comparator)
  Interventions: Drug: methyl aminolevulinate (MAL) and hexaminolevulinate (HAL)

INTERVENTIONS:
Drug: methyl aminolevulinate (MAL) and hexaminolevulinate (HAL) — MAL 1.2M, HAL 10mM and HAL 40mM solutions for 3 and 12 hours application

SUMMARY:
The study will determine the best drug (MAL or HAL) dosage for photodynamic therapy of cervical precancerous lesions (dysplasia) in women that are referred for conisation (surgery).

DETAILED DESCRIPTION:
Surgery (conisation) of precancerous cervical lesions (dysplasia) increase the risk of preterm deliveries in young women. Photodynamic therapy (PDT) is a selective, tissue preserving method that may become a good treatment option for these patients.

This study will explore topical application of methyl aminolevulinate (MAL) and hexaminolevulinate (HAL) of the cervix for photodynamic therapy using red light (630 nm). Different doses of MAL and HAL will be used with different application time, followed by illumination.

ELIGIBILITY:
Inclusion Criteria:

* Positive histology of CIN 1-3

Exclusion Criteria:

* Patients with endocervical lesions
* Patients with AGUS
* Patients with invasive disease
* Patients with porphyria
* Patients sensitive to MAL and HAL

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2006-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Lesion eradication | 6 months

SECONDARY OUTCOMES:
Eradication of lesion and HPV | 6 and 12 months
Safety assessment | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hillemanns, Md PhD, Principal Investigator — Hannover Medical School
Locations (2):
- Medizinische Hochschule Hannover, Department of Obstetrics and Gynecology, Hanover, Germany
- Ullevål University Hospital, Department of Obstetrics and Gynecology, Oslo, Norway